CLINICAL TRIAL: NCT02483975
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study of Once-daily Inhaled Fluticasone Furoate Inhalation Powder for Six Weeks on the Hypothalamic-pituitary-adrenocortical Axis of Children Aged 5-11 Years With Asthma
Brief Title: Effect of Fluticasone Furoate Inhalation Powder on the Hypothalamic-pituitary-adrenocortical Axis of Children Aged 5-11 Years With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 107118
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Asthma
Keywords: Fluticasone Furoate; Asthma; HPA axis; Children; Inhaled corticosteroid
MeSH Terms: conditions — Asthma | interventions — montelukast; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FF 50 mcg (Experimental): Subjects will receive by oral inhalation FF 50 mcg once daily in the morning via ELLIPTA for 42 days. Subjects will continue to receive oral montelukast once daily in the evening and may use albuterol/salbutamol inhalation aerosol as needed.
  Interventions: Drug: FF; Drug: Montelukast; Drug: Albuterol/Salbutamol
- Placebo (Placebo Comparator): Subjects will receive by oral inhalation placebo once daily in the morning via ELLIPTA for 42 days. Subjects will continue to receive oral montelukast once daily in the evening and may use albuterol/salbutamol inhalation aerosol as needed.
  Interventions: Drug: Placebo; Drug: Montelukast; Drug: Albuterol/Salbutamol

INTERVENTIONS:
Drug: FF — FF will be provided as a dry powder inhaler with 30 doses per device, each containing 50 mcg of FF as a dry white powder per blister, to be inhaled orally via ELLIPTA.
  Arms: FF 50 mcg
Drug: Placebo — Placebo will be provided as dry powder inhaler with 30 doses per device, each containing placebo as a dry white powder per blister, to be inhaled orally via ELLIPTA.
  Arms: Placebo
Drug: Montelukast — Montelukast will be provided as 4 mg and 5 mg chewable tablets.
Drug: Albuterol/Salbutamol — Albuterol/Salbutamol will be provided as inhalation aerosol.

SUMMARY:
Inhaled corticosteroids (ICS) have a number of known class effects including hypothalamic-pituitary-adrenocortical (HPA) axis suppression. Although the safety of inhaled Fluticasone Furoate (FF) on the HPA axis of adults and adolescent asthmatic patients has been established, it is important to assess the risk of suppression in children so as to establish whether this medicine can be safely used in this young population. This study aims to evaluate the effect of inhaled FF on the HPA axis of children 5-11 years of age (inclusive) with persistent asthma compared with placebo. Approximately 143 subjects will be enrolled. Subjects will enter a 7 to 14 day run-in period on oral montelukast 4 milligrams (mg) (5 year old subjects) or 5 mg (6-11 year old subjects) once daily. Eligible subjects will be randomized to receive once-daily FF inhalation powder 50 micrograms (mcg) or once-daily placebo inhalation powder in the morning via the ELLIPTA™ inhaler for 42 days. Subjects will continue to receive open label montelukast during the treatment period. All subjects will be provided albuterol/salbutamol inhalation aerosol, to use as needed to treat acute asthma symptoms throughout the study.

ELLIPTA is a registered trademark of the GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: Written informed consent from at least one parent/care giver and the accompanying informed assent from the subject (where the subject is able to provide assent) prior to admission to the study.

If applicable, subject must be able and willing to give assent to take part in the study according to the local requirement. The study investigator is accountable for determining a child's capacity to assent to participation in a research study, taking into consideration any standards set by the responsible Independent Ethics Committee (IEC)/Institutional Review Board (IRB).

Subject and their legal guardian understands that they must comply with study medication and study assessments.

* Age: 5-11 years (inclusive) at Visit 1.
* Weight: Subjects must weigh at least 17 kilograms (kg).
* Gender: Male and pre-menarchial female. Pre-menarchial females are defined as any female who has yet to begin menses.
* Diagnosis of asthma: Subjects must have a diagnosis of asthma documented in their medical history at least 6 months prior to Visit 1.
* Childhood Asthma Control Test (C-ACT): Subjects must have a C-ACT score of >19.
* Asthma Therapy Prior to Visit 1: Subjects are eligible if they have been using non-corticosteroid controller and/or short-acting beta2-agonist (SABA) bronchodilators alone for at least 4 weeks prior to Visit 1.
* Ability to use Dry Powder Inhalers: Subjects must demonstrate the ability to use the ELLIPTA inhaler under the supervision of their parents/caregiver.
* SABA: All subjects must be able to replace their current SABA treatment with albuterol/salbutamol aerosol inhaler at Visit 1 for use as needed for the duration of the study. Albuterol/salbutamol metered dose inhaler (MDI) will be administered with or without a spacer, to be used as determined by the investigator. The use or non-use of the spacer should be consistent for an individual subject throughout the study.
* Peak Flow Meter/Daily Diary Compliance: A subject must be able to use the study-provided peak flow meter and the subject/caregiver must be able to maintain the electronic diary record.

Exclusion Criteria:

* History of Life-Threatening Asthma: Subjects with a history of life-threatening asthma defined for this protocol as an asthma episode that required intubation, hypercapnea requiring non-invasive ventilatory support, respiratory arrest, hypoxic seizures or asthma-related syncopal episode(s).
* Asthma Exacerbation: Subjects with a history of asthma exacerbation requiring the use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days or a depot corticosteroid injection (within 3 months) or requiring hospitalization for asthma (within 6 months) prior to screening.
* Respiratory Infection: Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within 4 weeks of Visit 1 and led to a change in asthma management or in the opinion of the Investigator, expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Oropharyngeal Examination: A subject will not be eligible for the run-in if he/she has clinical visual evidence of candidiasis at Visit 1.
* Concurrent Disease: Any significant abnormality or medical condition identified at the screening medical assessment (including serious psychological disorder and congenital metabolic disorders) likely to interfere with the conduct of the study or affect the safety of the patient.
* Allergies/Intolerance:

Drug Allergy/Intolerance: Any adverse reaction including immediate or delayed hypersensitivity to any Leukotriene receptor antagonist (LTRA), or intranasal, inhaled, or systemic corticosteroid therapy. Known or suspected sensitivity/intolerance to the constituents of the powder inhaler (i.e. lactose) or montelukast (e.g. phenylalanine).

Milk Protein Allergy: History of severe milk protein allergy.

* Corticosteroid Use:

Administration of systemic, oral, or depot corticosteroids within 12 weeks of Visit 1 is prohibited and during the study.

Use of an ICS is prohibited during the 8 weeks prior to Visit 1 and during the study.

Use of intranasal corticosteroids is prohibited during the 4 weeks prior to Visit 1 and during the study.

Use of dermatological/topical corticosteroids during the 8 weeks prior to Visit 1 and during the study.

* Concomitant Medication: Use of prescription or over-the-counter medications that would significantly affect the course of asthma or the HPA axis system of subjects. In addition, use of potent cytochrome P450 3A4 (CYP3A4) inhibitors within 4 weeks of Visit 1 and during the study (e.g., Clarithromycin, atazanavir, indinavir, itraconazole, ketoconazole, nefazadone, nelfinavir; ritonavir; saquinavir; telithromycin, troleandomycin, voriconazole, mibefradil, cyclosporine).
* Tobacco/Marijuana Use: Present use of any tobacco or marijuana products.
* Affiliation with Investigator's Site: A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.
* Parental/ Guardian Factors: Parent or Guardian with a history of psychiatric disease, intellectual deficiency, substance abuse or other condition (e.g. inability to read, comprehend or write) which may affect: validity of consent to participate in the study, adequate supervision of the subject during the study, compliance of subject with study medication and study procedures (e.g. completion of daily diary, attending scheduled clinic visits) and subject safety and well-being.
* Children in Care: Children who are wards of the government or state are not eligible for participation in this study.
* Clinically significant obesity: Defined as greater than 98th percentile.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2015-10-09 (Actual); Primary Completion 2016-06-20 (Actual); Study Completion 2016-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- United States (11):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Alhambra, California
  - GSK Investigational Site, Costa Mesa, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Homestead, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Houston, Texas
- South Africa (3):
  - GSK Investigational Site, Middelburg, Mpumalanga
  - GSK Investigational Site, Panorama, Western Province
  - GSK Investigational Site, Bellville

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20329

REFERENCES:
- [Background] Bareille P, Tomkins S, Imber V, Tayob M, Dunn K, Mehta R, Khindri S. A randomized, double-blind, placebo-controlled, parallel-group study of once-daily inhaled fluticasone furoate on the hypothalamic-pituitary-adrenocortical axis of children with asthma. Allergy Asthma Clin Immunol. 2020 Feb 4;16:11. doi: 10.1186/s13223-020-0406-6. eCollection 2020. PMID 32042286

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants (par.) aged between 5 to 11 years with asthma were enrolled to either receive fluticasone furoate (FF) or placebo by inhalation through ELLIPTA for 6 weeks (wks) (42 days (D)). A total of 156 par. were screened, of which 111 par. were randomized in the study.
Pre-assignment Details: Par. receiving non-corticosteroid controller and/or short-acting beta 2-agonist (SABA) therapy were screened for the study. Par. went through a Run-in Period of 7 to 14 D before the 6 Wk Treatment Period.
Groups:
- Fluticasone Furoate 50 mcg: Par. received one inhalation, once daily of FF 50 microgram (mcg) in the morning via ELLIPTA inhaler for 6 wks. Par. also received open label montelukast throughout the treatment period and were supplied with albuterol/salbutamol inhalation aerosol to use as needed to treat acute asthma symptoms.
- Placebo: Par. received one inhalation, once daily of placebo in the morning via ELLIPTA inhaler for 6 wks. Par. also received open label montelukast throughout the treatment period and were supplied with albuterol/salbutamol inhalation aerosol to use as needed to treat acute asthma symptoms.
Period: Overall Study
Arm/Group | Fluticasone Furoate 50 mcg | Placebo
Started | 56 | 55
Completed | 54 | 53 (Subject reported as not completed due to AE was discontinued due to exacerbation, was not an AE/SAE)
Not Completed | 2 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fluticasone Furoate 50 mcg: Par. received one inhalation, once daily of FF 50 mcg in the morning via ELLIPTA inhaler for 6 wks. Par. also received open label montelukast throughout the treatment period and were supplied with albuterol/salbutamol inhalation aerosol to use as needed to treat acute asthma symptoms.
- Placebo: Par. received one inhalation, once daily of placebo in the morning via ELLIPTA inhaler for 6 wks. Participants also received open label montelukast throughout the treatment period and were supplied with albuterol/salbutamol inhalation aerosol to use as needed to treat acute asthma symptoms.
- Total: Total of all reporting groups
Arm/Group | Fluticasone Furoate 50 mcg | Placebo | Total
Number analyzed (Participants) | 56 | 55 | 111
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Overall study | 8.4 (1.97) | 8.4 (2.00) | 8.4 (1.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 30 | 50
  Male | 36 | 25 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 17 | 32
  Not Hispanic or Latino | 41 | 38 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 32 | 29 | 61
  White- White/Caucasian/European Heritage | 21 | 21 | 42
  Multiple-American Indian or Alaskan native & white | 0 | 1 | 1
  Multiple-East Asian Heritage & African American | 0 | 2 | 2
  Multiple- Asian-Japanese Heritage and White | 1 | 1 | 2
  Multiple- Black or African American and White | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Expressed as a Ratio) in 0-24 Hour Weighted Mean Serum Cortisol at the End of the Six Week Treatment Period (D 42) in Intention-to-treat (ITT) Population
Description: The blood samples for statistical analysis of serum cortisol (SC) endpoints were collected on D 0 and D 42 at the indicated time points. The weighted mean was calculated by dividing the area under the curve (AUC) over the 24-hour (hr) time period by the time period. Change from Baseline in 0-24 hr weighted mean SC was calculated as a ratio from Baseline defined as the SC weighted mean (0-24 hours) at Week 6 divided by the Baseline SC weighted mean (0-24 hours).The ratio from Baseline was loge transformed prior to analysis. The loge transformed ratios were compared between treatment groups as treatment ratios, using an analysis of covariance (ANCOVA) model, allowing for the effects of Baseline (loge transformed), age, sex and region. Treatment ratios for comparison was calculated by back-transforming the difference between the Least square (LS) means. Using the pooled estimate of variance, 95% Confidence Intervals (CIs) was calculated for the difference.
Time Frame: Baseline, D 0 (Pre-dose, 2hr, 4hr, 8hr, 12hr, 16hr and 24hr) and Day 42 (0hr, 2hr, 4hr, 8hr, 16hr and 24hr)
Population: ITT Population (pop) comprised of all randomized par. who received at least one dose of study medication. Randomized par. were assumed to have received study medication unless definitive evidence to the contrary exists. Par. with SC weighted mean (0-24 hr) calculated at Baseline and Week 6 were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Fluticasone Furoate 50 mcg | Placebo
Number analyzed (Participants) | 53 | 51
Ratio | 1.02 (46.71) | 1.01 (44.79)
Statistical Analysis 1: Comparison: Fluticasone Furoate 50 mcg vs Placebo; Test type: Non-Inferiority or Equivalence — Non inferiority was demonstrated if the lower limit of the two-sided 95% CI for the geometric mean ratio of each dose of fluticasone furoate 50 µg versus placebo was greater than 0.8; Least square Geometric Mean ratio = 0.92, 95% CI 2-sided [0.8040 to 1.0505]

2. Primary Outcome: Change From Baseline (Expressed as a Ratio) in 0-24 Hour Weighted Mean Serum Cortisol at the End of the Six Week Treatment Period (Day 42) in SC Population
Description: The blood samples for statistical analysis of serum cortisol (SC) endpoints were collected on D0 and D42 at indicated time points. The weighted mean was calculated by dividing the area under curve (AUC) over the 24-hr time period by time period. Change from Baseline in 0-24 hr weighted mean SC was calculated as a ratio from baseline defined as SC weighted mean (0-24 hrs) at Wk 6 divided by the baseline SC weighted mean (0-24 hrs). The ratio as treatment ratios, using an analysis of covariance (ANCOVA) model, allowing for the effects of baseline (loge transformed from baseline was loge transformed prior to analysis. The loge transformed ratios were compared between treatment groups), age, sex and region. Treatment ratios for comparison was calculated by back-transforming the difference between Least square (LS) means. Using the pooled estimate of variance, 95% CIs) was calculated for the difference.
Time Frame: Baseline, Day 0 (Predose, 2hr, 4hr, 8hr, 12hr, 16hr and 24hr) and Day 42 (0hr, 2hr, 4hr, 8hr, 16hr and 24hr)
Population: SC Population consisted of all par. in the ITT pop who did not have protocol violations that considered to affect the SC endpoint and whose serum samples were not considered to have confounding factors that would affect the interpretation of results. Par. with SC weighted mean (0-24 hr) calculated at baseline and Wk 6 were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Fluticasone Furoate 50 mcg | Placebo
Number analyzed (Participants) | 53 | 51
Ratio | 1.02 (47.16) | 1.00 (44.77)
Statistical Analysis 1: Comparison: Fluticasone Furoate 50 mcg vs Placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Least square Geometric Mean ratio = 0.93, 95% CI 2-sided [0.8096 to 1.0620]

3. Secondary Outcome: Change From Baseline (Expressed as a Ratio) in Area Under the Curve (AUC) 0-24 Hour Serum Cortisol at the End of the Six Week Treatment Period (Day 42).
Description: The blood samples for statistical analysis of area under the curve over the 24 hours (AUC 0-24 hours) endpoints were collected on Day 0 and Day 42 at the indicated time points. The AUC 0-24 hours was calculated using trapezoidal rule. Change from baseline in AUC 0-24 hour was calculated as a ratio from baseline defined as the AUC (0-24 hours) at Week 6 divided by the baseline AUC (0-24 hours) The ratio from baseline was loge transformed prior to analysis. The loge transformed ratios were compared between treatment groups as treatment ratios using an analysis of covariance (ANCOVA) model, allowing for the effects of baseline (loge transformed), age, sex and region. Treatment ratios for comparison was calculated by back-transforming the difference between the Least square (LS) means. Using the pooled estimate of variance, 95% Confidence Intervals (CIs) was calculated for the difference. Par. with SC weighted mean (0-24hr) calculated at baseline and Week 6 were analyzed
Time Frame: Baseline and Week Baseline, Day 0 (Predose, 2hr, 4hr, 8hr, 12hr, 16hr and 24hr) and Day 42 (0hr, 2hr, 4hr, 8hr, 16hr and 24hr)
Population: The SC population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Fluticasone Furoate 50 mcg | Placebo
Number analyzed (Participants) | 52 | 50
Ratio | 1.02 (47.11) | 1.00 (44.73)
Statistical Analysis 1: Comparison: Fluticasone Furoate 50 mcg vs Placebo; Test type: Superiority or Other; Least square Geometric Mean ratio = 0.93, 95% CI 2-sided [0.81 to 1.06]

4. Secondary Outcome: Change From Baseline (Expressed as a Ratio) in 24-hour Urinary Cortisol Excretion at the End of the Six Week Treatment Period (Day 42)
Description: The 24 hr urinary cortisol excretion was collected over a 24 hour period on Day 0 and Day 42. Change from baseline in 24- hr urinary cortisol excretion was calculated as a ratio from baseline defined as 24-hr urinary cortisol excretion at Week 6 divided by the baseline 24-hr urinary cortisol excretion. The ratio from baseline was loge transformed prior to analysis. The loge transformed ratio was compared between treatment groups using an analysis of covariance (ANCOVA) model, allowing for the effects of baseline (loge transformed), age, sex and region. Treatment ratios for comparison was calculated by back-transforming the difference between the Least square (LS) means. Using the pooled estimate of variance, 95% Confidence Intervals (CIs) was calculated for the difference. Participants with 24-hr urinary cortisol excretion at baseline and Week 6 were analyzed.
Time Frame: Baseline (Day 0) Day 42
Population: The Urinary Cortisol (UC) Population used consisted of all participants who did not have protocol violations that were considered to affect the urine cortisol endpoint and whose urine samples were not considered to have confounding factors that affect the interpretation of the results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Groups:
- Placebo: Par. received one inhalation, once daily of placebo in the morning via ELLIPTA inhaler for 6 wks. Par also received open label montelukast throughout the treatment period and were supplied with albuterol/salbutamol inhalation aerosol to use as needed to treat acute asthma symptoms.
Arm/Group | Fluticasone Furoate 50 mcg | Placebo
Number analyzed (Participants) | 51 | 50
Ratio | 0.69 (90.20) | 1.05 (123.86)
Statistical Analysis 1: Comparison: Fluticasone Furoate 50 mcg vs Placebo; Test type: Superiority or Other; Least square Geometric Mean ratio = 0.79, 95% CI 2-sided [0.61 to 1.03]

5. Secondary Outcome: Change From Baseline (Expressed as a Ratio) in 24-hour 6-beta Hydroxycortisol Excretion at the End of the Six Week Treatment Period (Day 42).
Description: The 24 hr urinary 6-beta hydroxycortisol excretion was collected over a 24 hour period on Day 0 and Day 42. Change from baseline in 24- hr urinary 6-beta hydroxycortisol excretion was calculated as a ratio from baseline defined as 24-hr urinary 6-beta hydroxycortisol excretion at Week 6 divided by the baseline 24-hr urinary 6-beta hydroxycortisol excretion. The ratio from baseline was loge transformed prior to analysis. The loge transformed ratio was compared between treatment groups using an analysis of covariance (ANCOVA) model, allowing for the effects of baseline (loge transformed), age, sex and region. Treatment ratios for comparison was calculated by back-transforming the difference between the Least square (LS) means. Using the pooled estimate of variance, 95% Confidence Intervals (CIs) was calculated for the difference. Participants with 24-hr urinary cortisol excretion at baseline and Week 6 were analyzed.
Time Frame: Baseline (Day 0) Day 42
Population: The UC Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Groups:
- Fluticasone Furoate 50 mcg: Participants received one inhalation, once daily of FF 50 mcg in the morning via ELLIPTA inhaler for 6 wks. Participants also received open label montelukast throughout the treatment period and were supplied with albuterol/salbutamol inhalation aerosol to use as needed to treat acute asthma symptoms.
- Placebo: Participants received one inhalation, once daily of placebo in the morning via ELLIPTA inhaler for 6 wks. Participants also received open label montelukast throughout the treatment period and were supplied with albuterol/salbutamol inhalation aerosol to use as needed to treat acute asthma symptoms.
Arm/Group | Fluticasone Furoate 50 mcg | Placebo
Number analyzed (Participants) | 50 | 49
Ratio | 0.78 (67.43) | 0.90 (65.54)
Statistical Analysis 1: Comparison: Fluticasone Furoate 50 mcg vs Placebo; Test type: Superiority or Other; Least square Geometric Mean ratio = 0.88, 95% CI 2-sided [0.72 to 1.07]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from participants up to 9 weeks.
Description: Safety analysis was based on Intent-to-Treat (ITT) population. Most frequent On-Treatment Non-serious AEs are reported. Most frequent is defined as >=3% (without rounding) in any treatment group. There were no fatal or non-fatal SAEs reported in the study.
Arm/Group | Fluticasone Furoate 50 mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/55
Other Adverse Events (participants affected / at risk) | 4/56 | 6/55
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Furoate 50 mcg (N=56) | Placebo (N=55)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Headache (Nervous system disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.